CLINICAL TRIAL: NCT06147765
Title: İnvestigation of the Relations Between Activity and Participation Levels, Social Skills and Behavior Levels of Children With Cerebral Palsy in Preschool Period and Parental Attitudes and Anxiety Levels
Brief Title: Relations Between Activity, Participation and Social Skills Levels of Preschool Cerebral Palsy and Parental Attitudes
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Melike Tanis, MELİKE TANIŞ, Hacettepe University
Other Study IDs: HacettepeU, MTanis
Record Dates: First submitted 2023-11-15; First posted 2023-11-28 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Cerebral Palsy (CP)
Keywords: Cerebral palsy; Physical activity; Social skills; Parent; Anxiety; attitude; Social participation
MeSH Terms: conditions — Cerebral Palsy; Motor Activity; Social Skills; Anxiety Disorders; Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cerebral palsy (CP) is a chronic condition which affects the development of motor function and posture, occurs as a result of injury or malformation in the developing central nervous system before, during or immediately after birth.

Depending on the health conditions accompanying motor and sensory problems of children with CP in the pre-school period, they are insufficient to be active in their daily lives, to play games, to spend time with their peers and to perform self-care activities.

In addition to care difficulties, economic difficulties, problems in reaching rehabilitation centers, many problems such as fear of their children's future, falling behind their peers, and who will take care of their children after them cause anxiety and stress for families. We can foresee that parenting attitudes may change in line with the anxiety and stress created by all these difficulties.

The investigator planned to do this study because we found that there is a need for studies examining the effects of the attitudes and anxiety levels of families of children with CP on children's activity and participation and social skills.

DETAILED DESCRIPTION:
in our study, the relationship between the attitudes and anxiety levels of parents with children with CP and the activity and participation levels of children will be examined. at the same time, it will be investigated whether there is a relationship between children's social skills and behaviors and physical activity and participation levels.

Eligibity Criteria:

cerebral palsy diagnosed 3-6 years Children or family who understand and speek Turkish language Children or family who know writing and reading Volunteer to join the study Going to pre-school education and/or special education and rehabilitation center for at least 3 months

Outcome Measures

Clinical classifications:

Gross Motor Function Classification System for classifying gross motor function levels Manuel ability classification system for classifying fine motor function levels Communication Function Classification System for classifying communication function levels Eating Drinking Abilities Classification System for classifying eating and drinking functions levels will be used

Physical Activity and Participation:

Gross Motor Function Measurement, Quality of Upper Extremity Skills Test, Bouchard Three-Day Physical Activity Record , Pediatric Evaluation of Disability Inventory, Child and Adolescent Scale of Participation will be used

Parental and Social Environment:

Parental Attitude Scale, Hospital Anxiety and Depression Scale, Preschool and Kindergarten Behavior Scale will be used.

ELIGIBILITY:
Inclusion Criteria:

* having been diagnosed with CP
* between the ages of 3-6
* parents/caregivers and those who speak Turkish
* their parents/caregivers are literate
* going to pre-school education and/or special education and rehabilitation center for at least 3 months
* those who agreed to participate in the study

Exclusion Criteria:

* different additional congenital and hereditary different disease that give system to CP
* children who have undergone any surgical procedure in the last 1 year

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Preschool children with CP
Sampling Method: Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2023-12-10 (Estimated); Primary Completion 2024-03-15 (Estimated); Study Completion 2024-05-15 (Estimated)

PRIMARY OUTCOMES:
Gross Motor Function Measurement | 10 minutes
  Children's motor ability will be assessed to investigate the correlations between the motor functions and orthosis used by child. The GMFM-88 consists of 88 items examining children's gross motor movements. Each item is scored between 0 and 3 points. The higher the child gets, the more successful the child is in gross motor functions.
Quality of Upper Extremity Skills Test | 10 minutes
  ıt was used to assess the function and quality of upper limb movements. This test has a total of 7 subdivisions, and the scoring of each section is calculated using a standardized formula. Each chapter is scored between 0-100 within itself. The first four section scores are used to calculate the total score. A high score indicates better the quality of the movement.
Bouchard Three-Day Physical Activity Record | at baseline
  ıt was used to measure daily energy expenditure in children and adolescents.ıt questions the activities that the children in two days during the week and one day on the weekend.
Pediatric Evaluation of Disability Inventory | 15 minutes
  It is a scale that evaluates the functional skills of the child and the help and manner of the caregiver, in which each part is evaluated separately as self-care, mobility and social function items.
Child and Adolescent Scale Of Participation (CASP) | 5 minutes
  Participation measurement The CASP consists of 20 ordinal-scaled items and four subsections: 1) Home Participation 2) Community Participation 3) School Participation and 4) Home and Community Living Activities The 20 items are rated on a four-point scale: Age Expected (Full participation) to Unable.

SECONDARY OUTCOMES:
Parental Attitude Scale | 5 minutes
  for measuring the child-rearing behaviors of the parents. This Likert-type scale was composed of four subscales including "Democratic", "Authoritarian", "Permissive" and "Protective"; and consisted of 46 items.
Hospital Anxiety and Depression Scale (HADS) | 5 minutes
  the scale is determining the levels of anxiety and depression that a person is experiencing.The HADS is a fourteen item scale that generates: Seven of the items relate to anxiety and seven relate to depression.
Preschool and Kindergarten Behavior Scales | 5 minutes
  the scale is a norm-referenced , standardized behavior rating scale designed to assess problem behaviors and social skills of children from ages 3 through 6 years.

CONTACTS AND LOCATIONS:
Overall Officials: Nezire Köse, Principal Investigator — Hacettepe University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Oskoui M, Coutinho F, Dykeman J, Jette N, Pringsheim T. An update on the prevalence of cerebral palsy: a systematic review and meta-analysis. Dev Med Child Neurol. 2013 Jun;55(6):509-19. doi: 10.1111/dmcn.12080. Epub 2013 Jan 24. PMID 23346889
- [Background] Shelly A, Davis E, Waters E, Mackinnon A, Reddihough D, Boyd R, Reid S, Graham HK. The relationship between quality of life and functioning for children with cerebral palsy. Dev Med Child Neurol. 2008 Mar;50(3):199-203. doi: 10.1111/j.1469-8749.2008.02031.x. Epub 2008 Jan 21. PMID 18215191
- [Background] Erkin G, Elhan AH, Aybay C, Sirzai H, Ozel S. Validity and reliability of the Turkish translation of the Pediatric Evaluation of Disability Inventory (PEDI). Disabil Rehabil. 2007 Aug 30;29(16):1271-9. doi: 10.1080/09638280600964307. PMID 17654002
- [Background] Eliasson AC, Krumlinde-Sundholm L, Rosblad B, Beckung E, Arner M, Ohrvall AM, Rosenbaum P. The Manual Ability Classification System (MACS) for children with cerebral palsy: scale development and evidence of validity and reliability. Dev Med Child Neurol. 2006 Jul;48(7):549-54. doi: 10.1017/S0012162206001162. PMID 16780622
- See also: The relationship between quality of life and functioning for children with cerebral palsy. — https://pubmed.ncbi.nlm.nih.gov/18215191/
- See also: Erkin G, Elhan AH, Aybay C, Sirzai H, Ozel S. Validity and reliability of the Turkish translation of the Pediatric Evaluation of Disability Inventory (PEDI). Disabil Rehabil. 2007 Aug 30;29(16):1271-9. — https://pubmed.ncbi.nlm.nih.gov/17654003/
- See also: Dammann O. Evidence-based child neurology. Dev Med Child Neurol. 2006 Jul;48(7):622-4. doi: 10.1017/S0012162206001307. PMID: 16780636. — https://pubmed.ncbi.nlm.nih.gov/16780622/